CLINICAL TRIAL: NCT04560465
Title: Efficacy of Tranexamic Acid in Reducing Myomectomy Associated Blood Loss in Federal Teaching Hospital Abakaliki
Acronym: AEFUTHA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alex Ekwueme Federal University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Olaleye Ayodele Adegbite, Dr, Alex Ekwueme Federal University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEFUTHA
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: To Determine Efficacy of Tranexamic Acid in Reducing Blood Loss During Myomectomy
Keywords: Tranexamic acid, Myomectomy, Blood loss, Gravimetric
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: two groups comprising of cases and control
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: Cases that had tranexamic acid infusion (Experimental): Group A had perioperative tranexamic acid infusion at the rate of 100mls per hour
  Interventions: Drug: Tranexamic acid
- Group B: Control (Placebo Comparator): control were given perioperative placebo at the rate of 100mls per hour
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — intravenous perioperative tranexamic acid was added into infusion of normal saline for the cases while placebo of intravenous water for injection was added into normal saline perioperatively for control

SUMMARY:
to determine safety and efficacy of Tranexamic Acid in reducing blood loss during Myomectomy in our institution.

DETAILED DESCRIPTION:
A double blinded randomized controlled trial in which cases were given 1000mg intravenous tranexamic acid into 1L of intravenous normal saline and control were given 10mls of placebo water for injection into same amount of intravenous fluid. outcome of both groups in terms of intraoperative blood loss, duration of surgery, postoperative packed cell volume and total blood loss with risk of blood transfusion were then determined.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women with symptomatic myomas women with no known contraindication to tranexamic acid

Exclusion Criteria:

* past history of thromboembolic disorder, ischaemic heart disease, malignancy or liver disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Average duration of surgery in each group | one year
  Average duration of Surgeries were calculated for each group
Mean intraoperative Blood loss | one year
  The mean intraoperative blood loss was calculated for both groups
Postoperative Haemoglobin concentration | one year
  Average Postoperative Haemoglobin concentration of both groups were determined

SECONDARY OUTCOMES:
Blood Transfusion | One year
  Risk of Blood Transfusion of both groups were determined

CONTACTS AND LOCATIONS:
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria

REFERENCES:
- [Derived] Olaleye AA, Adebayo JA, Eze JN, Ajah LO, Anikwe CC, Egede JO, Ebere CI. Efficacy of Tranexamic Acid in Reducing Myomectomy-Associated Blood Loss among Patients with Uterine Myomas at Federal Teaching Hospital Abakaliki: A Randomized Control Trial. Int J Reprod Med. 2024 Jan 18;2024:2794052. doi: 10.1155/2024/2794052. eCollection 2024. PMID 38283394